CLINICAL TRIAL: NCT04857970
Title: Impact of Routine Electronic Monitoring of Health-related Quality of Life on Care Relationship of Cancer Patients With Non-small Cell Lung Cancer, Locally Advanced or Metastatic, Systemic Treatment-naïve: a Randomized Trial
Brief Title: Routine Electronic Monitoring Of Quality Of Life -Poumon (REMOQOL-Poumon)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: University of Franche-Comté (Other); University of Burgundy (Other)
Responsible Party: Sponsor
Other Study IDs: P/2018/391
Record Dates: First submitted 2020-01-10; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer
Keywords: Cancer; Health-related quality of life; E-health; Patient-reported outcome
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Electronic HRQoL questionnaires with feedback to physicians: 40 patients allocated in this arm will answer HRQOL questionnaires using an electronic form in CHES Software. The HRQoL scores, presented as graphics, will be transmitted to physicians.
  Interventions: Other: Electronic HRQoL questionnaires with feedback to physicians
- Paper-pencil HRQoL questionnaires w.o. feedback to physician: 40 patients allocated in this arm will answer HRQOL questionnaires using "pencil-paper", without transmission of the HRQoL scores to physicians.
  Interventions: Other: Paper-pencil HRQoL questionnaires w.o. feedback to physicians

INTERVENTIONS:
Other: Electronic HRQoL questionnaires with feedback to physicians — Use of the CHES software for HRQoL collection and graphical display of the patients' HRQoL scores to physicians
  Groups: Electronic HRQoL questionnaires with feedback to physicians
Other: Paper-pencil HRQoL questionnaires w.o. feedback to physicians — Use of paper-pencil HRQoL questionnaires, the results of which are not presented to physicians
  Groups: Paper-pencil HRQoL questionnaires w.o. feedback to physician

SUMMARY:
Routine electronic monitoring of health-related quality of life (REMOQOL) consists of collecting HRQoL patients' data via an electronic device in order to provide these data to healthcare providers. Collected data could be used by professionals to personalize care through for instance, orientation towards personalized supportive care; assessment of toxicities related to treatments or adapted treatments.

The aim of this study is to investigate the impact of REMOQOL on the care relationship in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) who are naïve for systemic treatment. To do this, the investigators want to conduct a randomized trial at the Besançon University Hospital.

Several teams are collaborating on this project: Methodology and Quality of Life Unit in Oncology (UMQVC), pneumonology and medical oncology services of the Besançon University Hospital and psychology laboratories of Franche-Comté and Burgundy Universities.

The original aspects of this research are the particular interest in the care relationship between physicians and patients, also taking an interest in the physician's experience, the strong collaboration with researchers in psychology, the use of mixed quantitative and qualitative analysis techniques as well as the design of randomized study.

DETAILED DESCRIPTION:
REMOQOL-Poumon is an interventional, prospective, randomized study, conducted in Besançon University Hospital. Patients are randomized whether in the experimental arm or in the control arm. Intervention in experimental arm consists of administration of HRQoL questionnaires (QLQ-C30 & QLQ-LC13) using the CHES software (Computer-based Health Evaluation System) and presentation of the HRQoL scores to physicians via colored graphics.

In control arm, HRQoL questionnaires (QLQ-C30+LC13) are administered in a paper-pencil way, without transmission of results to physicians.

Patients are followed for four encounters with HRQoL collection. The primary outcome, measured with the AREP questionnaire, is assessed after those four encounters.

At the end of the follow-up, a semi-structured interview with a researcher in psychology and concerning the care relationship is proposed to a sub-cohort of patients (around ten patients in each arm).

After each encounter, physicians are asked to answer a questionnaire on viewing and use of HRQoL scores. Every physician will be interviewed on care relationship by a researcher in psychology.

ELIGIBILITY:
Inclusion Criteria for patients:

* Any patient diagnosed with locally advanced or metastatic non-small cell lung cancer
* Patients treated at University Hospital of Besançon
* No prior systemic therapy for cancer
* Males and Females, age ≥18 years old
* Patient able to complete the HRQoL questionnaires
* Patients who gave their informed consent to participate.

Inclusion Criteria for the sub cohort of patients undergoing the semi-structured interview with the researcher in psychology:

* Patients who realized 4 clinical encounters with collection of HRQoL
* For patients from experimental arm, the physician must have checked HRQoL results

Inclusion Criteria for physicians:

• Any physician treating patients included in the study REMOQOL-Poumon

Exclusion Criteria:

* Patients with tumor recurrence
* Patients receiving oral antineoplastic therapy for whom at least monthly follow-up is not feasible
* Patients with psychopathology or serious cognitive problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with locally advanced or metastatic non-small cell lung cancer + Physicians treating patients included in the study REMOQOL-Poumon
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
quality of care relationship, assessed for patients and physicians: AREP questionnaire | Month 3
  care relationship assessed with the AREP questionnaire. AREP is for "adjustment relationnel expérimenté perçu", which means experienced and perceived relational adjustment.

SECONDARY OUTCOMES:
Quality of care relationship, assessed for patients and physicians: semi-structured interviews | Month 24
  care relationship assessed with semi-structured interviews conducted by a researcher in psychology.
Descriptive characteristics: socio-demographic, clinic, treatments and HRQoL scores | Month 3
  Classical characteristics such as age at diagnosis, disease stage, type of treatments, HRQoL scores
Preferences and expectations in the care relationship, assessed for patients and physicians | Day 1
  preferences and expectations in the care relationship assessed with the Inventory of Expectations towards the care relationship (IARSS, for Inventaire d'Attentes envers la Relation Soignant-Soigné )
Acceptability of HRQoL collection | Month 24
  assessment of HRQoL collection considering usefulness, ease and user-friendliness
intention of use of REMOQOL | Month 24
Overall survival | Year 5
  Time from randomization to death from any cause, assessed at end of inclusion + 2 years
Progression-free survival | Year 5
  Time from randomization to disease progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Virginie WESTEEL, MD PhD, Principal Investigator — CHU de Besançon
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No